CLINICAL TRIAL: NCT03496194
Title: Anaesthesiological Involvement in Postoperative Pain Treatment - A Questionnaire Survey at Danish Hospitals
Brief Title: Anaesthesiological Involvement in Postoperative Pain Treatment
Status: Completed | Type: Observational
Sponsor: Zealand University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: ZUH
Record Dates: First submitted 2018-03-15; First posted 2018-04-12 (Actual); Last update posted 2021-11-18 (Actual); Status verified 2018-04

CONDITIONS: Pain, Postoperative; Anesthesia; Epidural Analgesia; Acute Pain
MeSH Terms: conditions — Pain, Postoperative; Acute Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Head of Post Anaesthesia Care Unit: The chief physician of PACUs at all Danish Anaesthesia departments will receive electronic survey on postoperative pain treatment

SUMMARY:
This study aims to investigate the current organization and management of postoperative pain in Denmark, especially for invasive pain treatment modalities (epidural infusions, PCA and regional blocks), in a national survey covering the activities in Danish Hospitals.

This study is an electronic questionnaire survey, that aim to describe and map the foundation for future developments within, and improvement of, postoperative pain management.

DETAILED DESCRIPTION:
Postoperative pain is one of the major challenges in postoperative care and several studies continue to demonstrate that postoperative pain is generally undertreated. A key focus for postoperative pain is to identify gold standards within procedure-specific pain treatment. However, results from single randomized trials do not per se lead to better treatment, as this requires both efforts within implementation of best evidence, quality control of efficacy, including efficacy on the individual level, and education of staff and physicians.

It has been suggested, that a way forward must include changes at the organizational level. For basic postoperative pain treatment, the major responsibility for planning and execution often rests on the surgical departments. For invasive pain treatment methods, e.g. epidural analgesia with continual infusion, patient controlled epidural analgesia (PCEA), patient controlled analgesia (PCA), and regional blocks, both single and continuing, this treatment is instituted at the departments of anaesthesia, but the responsibility for follow up is rarely described.

Generally, epidural analgesia is widely recommended because of superior benefits in reducing postoperative pain, pulmonal complications and surgical stress, as compared to systemic opioid treatment. However, epidural analgesia is not without complications especially not for abdominal and thoracic surgery. The accompanying unwanted motor blockade may delay recovery and recent studies question this treatment. Likewise, up to 20 % percent of patients will not receive adequate analgesia for the first 48 hours postoperative with this method. Finally, it is possible, that adverse effects and complications from epidural treatment are currently being underestimated, due to lack of routine monitoring and missing protocols.

Besides epidural analgesia, the use of Patient controlled analgesia (PCA), Patient controlled epidural analgesia (PCEA) and regional blocks have gained ground the last decades. With these techniques it might be possible to reduce overall opioid requirements. Nevertheless, a daily evaluation of benefits and harms of such analgesic techniques may be required to justify these treatment modalities. It is suggested, that regularly monitoring of invasive analgesic methods is of great concern when it comes to optimal postoperative pain management and reduction of adverse effects.

A structured organizational approach has the potential to improve benefit and harm of postoperative pain management. A number of studies argues that in order to obtain optimal postoperative pain treatment there need to be regular monitoring, and optimization of the analgesic regimens and techniques, preferably in a clinical setting with either an Acute Pain Service (APS) or a similar setup. With the decline of the use of APS's in Denmark it seems that the organization and management around postoperative pain treatment in general, and for invasive pain treatment methods in particular, needs to be investigated. As of today, it is not known how patients with such pain treatment are monitored and taken care of after leaving the post anaesthesia care unit, and where the responsibility for this pain treatment lies

ELIGIBILITY:
Inclusion Criteria:

* All departments of anesthesia with a PACU in Denmark

Exclusion Criteria:

* PACUs as part of day case surgery will be excluded

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Chief physicians for the postoperative care unit (PACU) at all Danish Departments of Anaesthesia
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2018-04-13 (Actual); Primary Completion 2018-05-05 (Actual); Study Completion 2018-06-06 (Actual)

PRIMARY OUTCOMES:
Proportion of hospitals, with a department of anesthesia, providing postoperative monitoring of epidural analgesia on postoperative day (POD) one. | From april 15th to may 1st 2018.
  The respondent will answer the question: "What invasive pain treatments are routinely inspected by the department of anesthesia" and choose from a list of options: "No", "Yes 1. POD", "Yes 2. POD", "Yes 3. POD" or "other": the respondent will specify.

SECONDARY OUTCOMES:
Size of hospital (number of beds) | From april 15th to may 1st 2018.
  Number of beds
Number of Post Anesthesia Care Units (PACU) | From april 15th to may 1st 2018.
  Number of PACU's
Size of PACU (number of beds) | From april 15th to may 1st 2018.
  Number of beds
Availability of a well defined acute pain unit with connected personnel | From april 15th to may 1st 2018.
  The respondent will choose "yes", "no" or "don't know"
Availability of a chronical pain unit/pain clinic | From april 15th to may 1st 2018.
  The respondent will choose "yes", "no" or "don't know"
Availability of a specialized pain unit for children | From april 15th to may 1st 2018.
  The respondent will choose "yes", "no" or "don't know"
Involvement of the department of anesthesia in inspection of patients with postoperative pain | From april 15th to may 1st 2018.
  The respondent will choose from a list of options: "On request from the ward", "Agreements on certain types of patients", "As a part of the work of the Acute Pain Service", "As part of the work of the chronical pain team", "We don't make inspections" or "Other": the respondent will specify.
Availability of a general protocol for postoperative pain in the PACU? | From april 15th to may 1st 2018.
  The respondent will choose "yes", "no" or "don't know"
Availability of a procedure specific protocol for postoperative pain | From april 15th to may 1st 2018.
  The respondent will choose "yes", "no" or "don't know"
Elaboration on the availability of a procedure specific protocol for postoperative pain between specialties | From april 15th to may 1st 2018.
  The respondent will choose "yes", "no", "not relevant for my department" or "don't know" for each specialty
Availability of protocols for perioperative management for patients with complicated pain issues and/or high opioid consumption | From april 15th to may 1st 2018.
  The respondent will choose "yes", "no" or "don't know"
Follow-up for patients with complicated pain issues after discharge from the hospital | From april 15th to may 1st 2018.
  The respondent will choose from a list of options: "Yes at the surgical department", "Yes at the multidisciplinary pain team/ chronical pain unit", "Yes at the local physician", "No follow-up", "Don't know" or "Other": the respondent will specify.
Type of invasive pain treatment offered | From april 15th to may 1st 2018.
  The respondent will choose from a list of options: "Epidural Pain Catheter", "PCEA", "PCA", "Regional Block (single shot)", "Regional Block (continual infusion)", "Regional Block (patient controlled bolus)", "Other": the respondent will specify og "No, none of the above"
Daily responsibility for follow-up/control of invasive pain treatment when the patients leave the PACU | From april 15th to may 1st 2018.
  The respondent will choose from a list of options: "Department of anesthesia", "The ward", "Don't know" or "Other": the respondent will specify
Routinely inspection by the department of anesthesia of the invasive pain treatment | From april 15th to may 1st 2018.
  The respondent will choose from a list of options:"No", "Yes 1. POD", "Yes 2. POD", "Yes 3. POD" or "other": the respondent will specify for each invasive pain treatment offered at the hospital.
Routinely inspection by the department of anesthesia of the invasive pain treatment with regards to involved personnel | From april 15th to may 1st 2018.
  The respondent will choose from a list of options: "Physician", "Nurse", "Acute pain team", "Chronical pain unit" or "Other": the respondent will specify.
Decisions on removal and duration of treatment with an epidural catheter | From april 15th to may 1st 2018.
  The respondent will choose from a list of options: "Department of anesthesia", "The ward", "Don't know" or "Other": the respondent will specify.
Involvement of the department of anesthesia in extension of the invasive pain treatment | From april 15th to may 1st 2018.
  The respondent will choose from a list of options: "Yes, every time", "Yes often", "Yes rarely", "No never" or "Don't know"
Participation of the department of anesthesia in other activities regarding postoperative pain treatment | From april 15th to may 1st 2018.
  The respondent will choose from a list of options: "Education in pain treatment", "Departmental quality assesment including guidelines and audits), "Implementation", "Research" or "Other": the respondent will specify.

CONTACTS AND LOCATIONS:
Overall Officials: Laura S Kruuse, Med.Student, Principal Investigator — Centre for Anaesthesiological research (CAR)
Locations (1):
- Centre for Anaesthesiological Research (CAR), Køge, Denmark

REFERENCES:
- [Background] Apfelbaum JL, Chen C, Mehta SS, Gan TJ. Postoperative pain experience: results from a national survey suggest postoperative pain continues to be undermanaged. Anesth Analg. 2003 Aug;97(2):534-540. doi: 10.1213/01.ANE.0000068822.10113.9E. PMID 12873949
- [Background] Mathiesen O, Thomsen BA, Kitter B, Dahl JB, Kehlet H. Need for improved treatment of postoperative pain. Dan Med J. 2012 Apr;59(4):A4401. PMID 22459715
- [Background] White PF, Kehlet H. Improving postoperative pain management: what are the unresolved issues? Anesthesiology. 2010 Jan;112(1):220-5. doi: 10.1097/ALN.0b013e3181c6316e. No abstract available. PMID 20010418
- [Background] Ready LB, Oden R, Chadwick HS, Benedetti C, Rooke GA, Caplan R, Wild LM. Development of an anesthesiology-based postoperative pain management service. Anesthesiology. 1988 Jan;68(1):100-6. doi: 10.1097/00000542-198801000-00016. No abstract available. PMID 3337359
- [Background] Nielsen PR, Christensen PA, Meyhoff CS, Werner MU. Post-operative pain treatment in Denmark from 2000 to 2009: a nationwide sequential survey on organizational aspects. Acta Anaesthesiol Scand. 2012 Jul;56(6):686-94. doi: 10.1111/j.1399-6576.2012.02662.x. Epub 2012 Mar 5. PMID 22385392
- [Background] Rawal N. Current issues in postoperative pain management. Eur J Anaesthesiol. 2016 Mar;33(3):160-71. doi: 10.1097/EJA.0000000000000366. PMID 26509324
- [Background] Rawal N. Epidural technique for postoperative pain: gold standard no more? Reg Anesth Pain Med. 2012 May-Jun;37(3):310-7. doi: 10.1097/AAP.0b013e31825735c6. PMID 22531384
- [Background] Burstal R, Wegener F, Hayes C, Lantry G. Epidural analgesia: prospective audit of 1062 patients. Anaesth Intensive Care. 1998 Apr;26(2):165-72. doi: 10.1177/0310057X9802600206. PMID 9564395
- [Background] Breivik H, Norum HM. [Regional analgesia--risks and benefits]. Tidsskr Nor Laegeforen. 2010 Feb 25;130(4):392-7. doi: 10.4045/tidsskr.08.0220. Norwegian. PMID 20220867
- [Background] Golster M. Seven years of patient-controlled epidural analgesia in a Swedish hospital: a prospective survey. Eur J Anaesthesiol. 2014 Nov;31(11):589-96. doi: 10.1097/EJA.0000000000000105. PMID 24922048
- [Background] Duncan F. Prospective observational study of postoperative epidural analgesia for major abdominal surgery. J Clin Nurs. 2011 Jul;20(13-14):1870-9. doi: 10.1111/j.1365-2702.2011.03752.x. Epub 2011 May 25. PMID 21615577